CLINICAL TRIAL: NCT00455819
Title: Home Treatment of Patients With Pulmonary Embolism Based on Pro-BNP Levels
Brief Title: Home Treatment of Patients With Pulmonary Embolism Based on Pro-Brain Natriuretic Peptide (BNP) Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: Diakonessenhuis, Utrecht (Other); Groene Hart Ziekenhuis (Other); Reinier de Graaf Groep (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTME/VL-06.12; HOME
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; pro-BNP; home treatment
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: home treatment

SUMMARY:
The aim of this study is to investigate the safety of treatment of pulmonary embolism in an outpatient setting based on normal pro-BNP levels. The mortality rate and the incidence of hemodynamic instability as well as major bleeding and recurrent venous thromboembolism (VTE) in the outpatient group will be studied.

DETAILED DESCRIPTION:
Pulmonary embolism is a major health problem. Because of risk for early hemodynamic instability and mortality, all patients with a recently diagnosed pulmonary embolism are treated in hospital. The clinical course of most patients is without complications. In practice most of the patients are only waiting in hospital in a good, clinical stable condition until their INR range is stable.

This prospective management study is to investigate the safety of treatment of pulmonary embolism in an outpatient setting based on normal pro-BNP levels (< 500 pg/ml). The incidence of complications due to the pulmonary embolism or its treatment will be followed during the first ten days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* outpatient with a pulmonary embolism, confirmed by locally approved guidelines
* aged 18 years and above
* written informed consent

Exclusion Criteria:

* hemodynamic or respiratory instability defined as one of the following; hypotension RR systolic< 90 mmHg,pulse rate> 100 bpm, need for oxygen therapy to maintain oxygen saturation above 90 %, collapse
* illness unrelated to PE for which the patient would require hospitalization
* pain requiring intravenous narcotics
* thrombolysis
* active bleeding or thrombopathy
* pregnancy
* in hospital patients
* physical or psychiatric inability for home treatment
* no support system at home renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Mortality rate due to pulmonary embolism or its treatment during a period of ten days in the outpatient group

SECONDARY OUTCOMES:
Rate of re-admission due to pulmonary embolism or its treatment in the outpatient group: hemodynamic instability, major bleeding, recurrence of venous thromboembolism

CONTACTS AND LOCATIONS:
Overall Officials: Douwe H Biesma, D.H., Study Director — St. Antonius Hospital
Locations (2):
- Netherlands (2):
  - St Antonius Hospital, Nieuwegein
  - Mesos Medical Centre, Utrecht

REFERENCES:
- [Derived] Agterof MJ, Schutgens RE, Snijder RJ, Epping G, Peltenburg HG, Posthuma EF, Hardeman JA, van der Griend R, Koster T, Prins MH, Biesma DH. Out of hospital treatment of acute pulmonary embolism in patients with a low NT-proBNP level. J Thromb Haemost. 2010 Jun;8(6):1235-41. doi: 10.1111/j.1538-7836.2010.03831.x. Epub 2010 Mar 3. PMID 20230418